CLINICAL TRIAL: NCT01491763
Title: Chemotherapy and Imatinib in Young Adults With Acute Lymphoblastic Leukemia Ph (BCR-ABL) POSITIVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL Ph-2008
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia Ph Positive
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imatinib — 600 mg p.o. from day 1 until consolidation

SUMMARY:
20-25% of patients over 15 years with acute lymphoblastic leukemia (ALL) have the Philadelphia chromosome or BCR-ABL rearrangement. Traditionally, intensive chemotherapy followed by hematopoietic stem cell transplantation (HSCT) have formed the basis allogeneic treatment of this disease, but the results have been poor (60-75% complete remissions-RC-and probability of long-term survival less than 20%). The effectiveness of imatinib for hematologic responses in patients with Ph + (observed in phase I and II) led to its use in phase III trials in combination with chemotherapy. They saw a chance of obtaining the RC above 90%, with acceptable toxicity, a molecular response rate (MR) of 40-50%, and prolonged follow-up studies, a probability of disease-free survival (DFS ) of 30-50%, significantly higher than historical controls with the same chemotherapy without imatinib. This led to the approval of imatinib by the rating agencies in the U.S., Europe and Japan as a treatment for Ph + in combination with chemotherapy.

Of the studies that led to the approval of this indication for imatinib, and other incurred after, the following conclusions can be drawn:

There is no specific pattern of combination of imatinib (at doses of 600 mg / day, po) and chemotherapy. However, when compared with concomitant alternating with the first achieved a higher rate of RM at the end of induction, although this did not influence DFS.

In studies in elderly patients has achieved a high CR rate (almost 100% in all series), only imatinib and glucocorticoids, suggesting that an attenuated induction may be sufficient to achieve CR in young patients with minimal toxicity, which further compromises the administration of treatment and allow for an allogeneic HSCT with minimal toxic load possible.

Although there is no consensus on the indication of allogeneic HSCT in first CR when given imatinib associated with intensive chemotherapy is an option that is done in most studies.

The allogeneic HSCT is most effective when carried out in complete molecular response to or greater than when there is more residual disease. However, the impact of MRI to obtain early (after induction) on survival is not clear. So far-reaching goal is to make the TPH in complete molecular response situation or greater.

The relapse of the disease at the molecular level is still short-term (less than 3 months) of hematological relapse. This implies the need for frequent monitoring of residual disease (ER) The frequency of relapse post HSCT is high (around 30%), raising the need for any post HSCT treatment, including imatinib included. Are currently ongoing clinical trials comparing the systematic administration of imatinib after administration TPH face is detected only when ER.

The applicability of the administration of imatinib after HSCT is limited by toxicity related to the procedure of TPH, is making frequent dose reduction or discontinuation.

Therefore, a reasonable approximation treatment of Ph + outside the context of a clinical trial is to get as many molecular responses before allogeneic HSCT in a position to make the same MRI complete or greater. After TPH, must be very close monitoring of the ER, and imatinib is administered as soon as you notice the loss of molecular response.

In patients who can not make an allogeneic HSCT for lack of histocompatible donor or contraindications for its realization it is recommended imatinib and chemotherapy, although there are studies that have undergone an autologous HSCT, followed or not treatment "maintenance" with imatinib. The low toxicity of autologous HSCT and no effect of graft versus leukemia are strongly recommended the administration of maintenance therapy with imatinib combined with chemotherapy or not.

DETAILED DESCRIPTION:
Induction Chemotherapy

* Vincristine (VCR): 1.5 mg/m2 (maximum dose 2 mg) iv days 1, 8, 15 and 22
* daunorubicin (DNR) 45 mg/m2 i.v. days 1, 8, 15 and 22
* Prednisone (PDN): 60 mg/m2 per day, i.v. or p.o., days 1-27
* Imatinib 600 mg p.o. from day 1 until the beginning of the consolidation. Important Note: The administration of imatinib be initiated as soon as the outcome of cytogenetic and molecular study, which will be known under normal conditions during prophase consolidation

Patients should be in RC and shall be a minimum of 2 weeks of finding it. Patients did not discontinue treatment with imatinib during this period. Minimum counts to start the consolidation are: neutrophils> 1x109 / L and platelets> 100x109 / L.

* Mercaptopurine (MP) 50 mg/m2, p.o. days 1 to 7, 28 to 35 and 56 to 63
* MTX: 1.5 g/m2, i.v. continuous infusion for 24 hours on days 1, 28 and 56.
* VP-16: 100 mg/m2 every 12 hours, i.v. (1 hour infusion) on days 14 and 42
* ARA-C: 1000 mg/m2 every 12 hours, i.v. (3-hour infusion) days 14-15 and 42-43
* triple intrathecal treatment days 1, 28 and 56
* Imatinib 600 mg / d po, from day 1 to 15 days before the TPH.

During consolidation therapy is recommended in primary prophylaxis with G-CSF or found neutropenia (<0.5 x109 / L). This factor was administered daily until the neutrophil count is > 1x109 / L in two consecutive measurements. Alternatively, PEG-filgrastim can be used (eg 16 and 44), at the discretion of each center

Allogenic THP or Autologous TPH

ELIGIBILITY:
Inclusion Criteria:

* Patients with Ph (BCR/ABL) positive de novo < 55 years old (it is advisable to include patients over 55 years LAL07OPH protocol).
* Performance status 0-2 (Appendix B) may include patients with performance status > 2 attributable to LAL.
* Patients without functional impairment of organs: liver function: total bilirubin, AST, ALT, alfa-GT and alkaline phosphatase less than 3 times the upper limit of normal laboratory renal function: serum creatinine < 2 mg/dL or clearance creatinine > 30 ml/min (except renal function attributable to LAL) cardiac function (Appendix B) normal: ventricular EF > 50%, absence of severe chronic respiratory disease. In the event that alterations are secondary to the disease is at the discretion of the investigator to determine if the patient can be included in the trial.

Exclusion Criteria:

* Any other variety of LAL
* Patients with a history of coronary artery disease, valvular or hypertensive heart disease
* Patients with chronic liver disease
* Patients with chronic respiratory failure
* Renal failure not due to LAL
* Patients with positive HIV status
* No serious neurological abnormalities due to LAL
* Impact on overall severe (grade 3 or 4 of the WHO scale) not attributable to the LAL
* Pregnant or breastfeeding
* initial blast crisis CML

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of number of complete response | 1 year

CONTACTS AND LOCATIONS:
Locations (74):
- Spain (74):
  - H. Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Germans Trias i Pujol and all Hospital Pethema, Badalona, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital general de Castellón, Castelló, Castellón
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General de Albacete, Albacete
  - Hospital de Alcorcón, Alcorcón
  - Hospital General de Alicante., Alicante
  - Hospital de Cabueñes, Asturias
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital Clínico y Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital de la santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Duran i Reynals - ICO L'Hospitalet, Barcelona
  - Basurtuko Ospitalea, Basurto
  - Complejo Hospitalario de Cáceres, Cáceres
  - Complejo Hospitalario Reina Sofía, Córdoba
  - Area Hospitalaria Juan Ramón Jimenez, Huelva
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital del SAS de Jerez de la Frontera, Jerez de la Frontera
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Arnau de Vilanova, Lleida
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Clínica La Concepción, Madrid
  - Clínica Puerta de Hierro, Madrid
  - Hospital 12 de Octubre. Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital de Madrid, S.A.- Norte Hospital General, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Princcipe de Asturias, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Carlos Haya, Málaga
  - Hospital de Mérida, Mérida
  - Hospital General Univeristario Morales Messeguer, Murcia
  - Hospital Sta. Maria del Rosell, Murcia
  - Hospital del Río Carrión, Palencia
  - Hospital de Gran Canaria Doctor Negrín, Palma de Gran Canaria
  - Clínica Universitaria de Navarra, Pamplona
  - Hospital de Montecelo, Pontevedra
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario, Salamanca
  - Hospital de Donostia, San Sebastián
  - Hoaspital Marqués de Valdecilla, Santander
  - Hospital General de Segovia, Segovia
  - Complejo Hospitalario Regional Virgen del Rocío, Seville
  - Hospital Joan XIII de, Tarragona
  - Hospital Joan XXIII, Tarragona
  - Hospital Clínico de Valencia., Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Clínico Universitario, Valencia
  - Hospital Clínic, Valencia
  - Hospital Dr Pesset, Valencia
  - Hospital La Fe, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Xeral-Cies, Vigo
  - Hospital do Meixoeiro, Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Clínico Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Ribera JM, Garcia O, Moreno MJ, Barba P, Garcia-Cadenas I, Mercadal S, Montesinos P, Barrios M, Gonzalez-Campos J, Martinez-Carballeira D, Gil C, Ribera J, Vives S, Novo A, Cervera M, Serrano J, Lavilla E, Abella E, Tormo M, Amigo ML, Artola MT, Genesca E, Bravo P, Garcia-Belmonte D, Garcia-Guinon A, Hernandez-Rivas JM, Feliu E; PETHEMA Group of the Spanish Society of Hematology. Incidence and outcome after first molecular versus overt recurrence in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia included in the ALL Ph08 trial from the Spanish PETHEMA Group. Cancer. 2019 Aug 15;125(16):2810-2817. doi: 10.1002/cncr.32156. Epub 2019 Apr 23. PMID 31012967
- See also: Pethema Foundation — https://www.fundacionpethema.es/